CLINICAL TRIAL: NCT02122887
Title: Peace-Building Interventions for Israeli and Palestinian Youth: Effects on Biological and Behavioral Markers of Empathy, Prejudice, and Dialogue
Brief Title: Peace-Building Interventions for Israeli and Palestinian Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Moran Influs, research manager, Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BIU901305
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: jewish, arab, israel, teenagers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): no intervention for 3 months
- experimental group (Experimental): Peace-Building Intervention Process- The intervention process consists of eight sessions and adheres to a manualized protocol that we developed. Each session lasts 120 minutes.
  Interventions: Behavioral: Peace-Building Intervention Process

INTERVENTIONS:
Behavioral: Peace-Building Intervention Process — The eight sessions include (1) presentation of the self to others members (2) getting familiar with the other culture (3) what is a conflict - how do conflicts come about, what are adaptive and non-adaptive modes of resolving conflict (4) getting to know the "Other" - preconceived notions about the other side (5) on dialogue- what is dialogue, can dialogue offer means for conflict resolution, what are the benefits of dialogue to inter-cultural and inter-racial conflicts, (6) empathy, generosity, and kindness (7) wrapping up - hopes for the future at the personal and community levels, practical suggestions (8) goodbye and summary - what have we learned ,"gift giving", summary of process by group leaders.
  Arms: experimental group

SUMMARY:
The investigators expect an intervention that focuses on actual dialogue and familiarity with members of the other culture, discussion of empathy, generosity, and kindness, and focus on adaptive and reciprocal modes of conflict resolution will alter both physiological, behavioral, and mental response to the pain of the other, increase empathy, and reduce hostility.

DETAILED DESCRIPTION:
We hypothesized that the intervention will impact perspective taking (PT) on the national conflict, reducing the tendency to view justice only on one's side. Such increase in PT would initiate a chain leading to greater behavioral empathy.

Second, we hypothesize that change in oxytocin (OT) levels and empathic behavior (less withdrawal and tension and more synchrony) would be impacted by the intervention and the degree to which it altered youth PT on the conflict.

Finally, we suggest a 3-path model charting the multi-dimensional pathways leading to behavioral empathy toward outgroup member. First, individual differences in OT functionality will shape empathy so that youth with higher OT levels at pre-intervention and greater PT will show more empathic dialogue at post-intervention. Second, dispositional cognitive empathy, as tested by the Interpersonal Reactivity Index questioner (IRI), at pre-intervention will predict higher behavioral empathy at T2, both directly and as mediated by reduction in ethnocentric attitudes following the intervention. Finally, we hypothesize that the intervention will influence empathy by initiating a chain that begins with increasing PT, which, in turn, will lead to reduction in tension during interaction with outgroup, and culminating in greater empathy during face-to-face encounters

ELIGIBILITY:
Inclusion Criteria:

* jewish israeli
* arab israeli
* lives in the center of israel
* both parents agree to participation

Exclusion Criteria:

* no mental disorder
* no neurological-developmental disorder

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moran Influs, MA, Principal Investigator — Bar Ilan University, Ramat Gan, Israel
Locations (1):
- Bar Ilan University, Ramat Gan, Israel

REFERENCES:
- [Derived] Influs M, Masalha S, Zagoory-Shaon O, Feldman R. Dialogue intervention to youth amidst intractable conflict attenuates stress response to outgroup. Horm Behav. 2019 Apr;110:68-76. doi: 10.1016/j.yhbeh.2019.02.013. Epub 2019 Mar 9. PMID 30807738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 60 | 41
Completed | 40 | 39
Not Completed | 20 | 2
Not completed — Withdrawal by Subject | 20 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.43 (.79) | 16.64 (.74) | 16.54 (.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 18 | 17 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ethnicity: Jewish | 20 | 19 | 39
  ethnicity: Arab | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  Israel | 40 | 39 | 79
Empathy (IRI-INTERPERSONAL REACTIVITY INDEX ) [Mean (Standard Deviation); unit: units on a scale] — Interpersonal Reactivity Index (IRI) (Davis, 1980) The instrument contains four seven-item subscales (as 7 is the highest and 1 is the lowest), taping facets of empathy: 1) Empathic concern 2) Perspective taking 3) Personal distress scale 4) Fantasy scale measures the tendency to imaginatively transpose oneself into fictional situations. We used only the perspective-taking scale, assessing tendency to spontaneously adopt viewpoints of others in everyday life, as relevant to our research. Scores for each subscale can ranges from 7 (for low empathy) to 49 (for the most empathic person). Population: 1 participant data was lost
  units on a scale
    number analyzed (Participants) | 40 | 38 | 78
    (all) | 17.71 (2.06) | 18.96 (2.83) | 18.63 (3.83)
Ethnocentrism [Mean (Standard Deviation); unit: units on a scale] — Ethnocentrism Scale- This Revised Ethnocentrism Scale contains 22 items with 15 scored and 7 mark balance between numbers of statements regarding subject's perception of other cultures in comparison to own culture. Each Item is scored on a scale from 1 to 5, 1 is strongly disagree and 5 is strongly agree. Total score for this scale is 15 at the lowest, for someone very open to other cultures, and 75 at the highest, for the most ethnocentric person.
  units on a scale | 35.2 (8.83) | 33.89 (10.61) | 34.56 (9.71)

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Assessment of Dialogue
Description: Interactions were coded with the "Coding Interactive Behavior" (CIB) manual (Feldman, 1998), adolescent version. This version of the CIB is composed of 32 codes rated on a scale of 1 to 5, as higher score mean a better outcome. The Two following constructs were used: A personal measure of "Behavioral Empathy" - an average of the following CIB codes: expressing empathy, acknowledging other's communication, elaborating other's topics and ideas, maintaining positive affect, maintaining visual, and give-and-receive reciprocity and Dyadic Tension - averaged codes; displaying a tense, anxious, and uneasy behavior, fear, and constriction of communicative output and social behavior.
Time Frame: trail 1-baseline
Population: All participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 40 | 39
units on a scale
  Behavioral Empathy | 3.07 (.81) | 3.21 (.98)
  Dyadic Tension | 2.26 (1.04) | 2.23 (1.14)

2. Primary Outcome: Hormonal Assays- Oxytocin
Description: Three saliva samples were collected using Salivettes® at baseline, following interaction, and ten minutes after end and averaged. All samples were then stored at -20°C. Salivette were treated as following: centrifuged twice, at 4°C at 1500 x g for 30 minutes, aliquoted and lyophilized over few days- to concentrate by 4 times. The dry samples were reconstructed in the assay buffer immediately before analysis using an oxytocin enzyme immunoassay commercial kit (ENZO, NY). The assay preformed according the kit's instruction. The concentration of oxytocin was calculated using MatLab-7
Time Frame: trail 1- baseline
Population: Some participants didn't have a measure due to insufficient saliva
Measure: Mean (Standard Deviation); unit: picogram/ml
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 33 | 39
picogram/ml | 44.08 (26.67) | 49.93 (34.41)

3. Primary Outcome: PT (Perspective-taking)
Description: Participants were interviewed individually on their attitudes towards the Israeli-Palestinian conflict. Perspective-taking (PT), addressed the degree to which adolescents thought justice was solely on their side and the other side is totally wrong, aggressive, and vicious compared to the ability to see some justice on both sides. Participants received binary score for PT, as 1 is some ability to see justice on the other side, and 0 is seeing justice only in own side.
Time Frame: trail 1-baseline
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 40 | 39
Participants
  justice is solely on our side | 21 | 21
  There is some justice in the other side | 19 | 18

4. Secondary Outcome: Behavioral Assessment of Dialogue
Description: as for outcome 1
Time Frame: trail 2- 3 months after trail 1
Population: Control group had few missing values due to problems in the interaction videos that didn't allow data analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 36 | 39
units on a scale
  Behavioral Empathy | 3.33 (.81) | 3.29 (.79)
  Dyadic Tension | 1.8 (.90) | 1.84 (.89)

5. Secondary Outcome: Hormonal Assays-Oxytocin
Description: as for outcome 2
Time Frame: trail 2- 3 months after trail1
Population: Some participants didn't have a measure due to insufficient saliva
Measure: Mean (Standard Deviation); unit: picogram/ml
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 38 | 38
picogram/ml | 40.03 (57.43) | 43.42 (35.34)

6. Secondary Outcome: Changes in PT (Perspective-taking) After Intervention
Description: Participants were interviewed individually on their attitudes towards the Israeli-Palestinian conflict. Perspective-taking (PT), addressed the degree to which adolescents thought justice was solely on their side and the other side is totally wrong, aggressive, and vicious compared to the ability to see some justice on both sides. Participants received binary score for PT.
Time Frame: trail 2- 3 months after trail 1
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 40 | 39
Participants
  justice is solely on our side | 16 | 24
  There is some justice in the other side | 24 | 15
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; we hypothesised that following intervention, those undergoing intervention will be more likely to see justice on both sides, compared to control group; Test type: Other — χ² (1) =4.57, Cramer's V=.24; p < 0.05, Chi-squared

7. Secondary Outcome: Changes in Tension as a Function of Perspective-taking and Group
Description: Perspective-taking (PT), addressed the degree to which adolescents thought justice was solely on their side compared to the ability to see some justice on both sides. Participants received binary score for PT and were divided to high vs low PT groups accordingly.
  We compared participants' tension levels, according to level of PT and group (intervention or control). Interactions were coded with the "Coding Interactive Behavior" (CIB) manual (Feldman, 1998), adolescent version. This version of the CIB is composed of 32 codes rated on a scale of 1 to 5, as higher score means a better outcome. Dyadic Tension is the averaged codes; displaying a tense, anxious, and uneasy behavior, fear, and constriction of communicative output and social behavior.
Time Frame: trail 2- 3 months after trail1
Population: All participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 40 | 39
units on a scale
  High Perspective-taking: number analyzed (Participants) | 19 | 18
  High Perspective-taking | 2.13 (0.81) | 2.18 (1.01)
  Low Perspective-taking: number analyzed (Participants) | 21 | 21
  Low Perspective-taking | 2.67 (0.85) | 2.39 (1.01)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; Test type: Equivalence — we compared participants levels of tension (in their interaction with an outgroup member in trail 2) in an interaction test between perspective-taking levels and group; p > 0.05, ANOVA; df=1; Mean Difference (Final Values) = .65

8. Secondary Outcome: Changes in Empathy as a Function of Perspective Taking
Description: Perspective-taking (PT), addressed the degree to which adolescents thought justice was solely on their side compared to the ability to see some justice on both sides. Participants received binary score for PT and were divided to high vs low PT groups accordingly.
  We compared participants' behavioral empathy levels. Interactions were coded with the "Coding Interactive Behavior" (CIB) manual (Feldman, 1998), adolescent version. This version of the CIB is composed of 32 codes rated on a scale of 1 to 5, as higher score means a better outcome. "Behavioral Empathy" is the average of the following CIB codes: expressing empathy, acknowledging other's communication, elaborating other's topics and ideas, maintaining positive affect, maintaining visual, and give-and-receive reciprocity
Time Frame: trail 2- 3 months after trail 1
Population: All participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 40 | 39
units on a scale
  High Perspective-taking: number analyzed (Participants) | 19 | 18
  High Perspective-taking | 1.58 (0.83) | 1.43 (0.86)
  Low Perspective-taking: number analyzed (Participants) | 21 | 21
  Low Perspective-taking | 1.38 (0.63) | 1.16 (0.39)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; Test type: Equivalence — we compared participants levels of empathy (in their interaction with an outgroup member in trail 2) in an interaction test between perspective-taking levels and group; p > 0.05, ANOVA; Mean Difference (Final Values) = 0.04

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Groups:
- no Intervention for 3 Months: This group did not received any intervention
Arm/Group | no Intervention for 3 Months | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Larger numbers are required before generalizations can be made. Participants had inters on resolving the conflict, enrolled from their own free will.

The intervention group got no other intervention. We measured peripheral, not central Oxytocin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes